CLINICAL TRIAL: NCT05555368
Title: Turkish Validity and Reliability of the Recovery Scale QoR-15
Acronym: Qor-15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, ümmühan kılıç, Principal Investigator, Ondokuz Mayıs University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Recovery Scale
Record Dates: First submitted 2022-08-22; First posted 2022-09-26 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single group (Other): The Qo0R-15 scale will be administered to 150 patients.
  Interventions: Other: Quality of Recovery Score

INTERVENTIONS:
Other: Quality of Recovery Score — Descriptive
  Other Names: Turkish validity and reliability

SUMMARY:
It is adapted and encouraged to a point to improve their quality of intervention for the purpose of the research.

DETAILED DESCRIPTION:
This research was conducted as a methodological and descriptive study to evaluate the psychometric properties of the "Quality of Recovery Score" in patients who had surgery. The study was carried out with the participation of 150 patients over the age of 18 who were operated under general anesthesia in Samsun Training and Research Hospital between 8.11.2021 and 3.01.2022.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* operated under general anesthesia

Exclusion Criteria:

* non-operative under general anesthesia
* under 18 years old

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
The Turkish validity of the QoR-15 version of the Quality of Healing Scale | 6 mounth
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Ümmühan Kılıç, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with anyone.